CLINICAL TRIAL: NCT05680584
Title: Comparison Between the Effect of Oral Melatonin and Hydroxyzine for Preventing Preoperative Anxiety in Pediatric Patients Undergoing Adenotonsillectomy
Brief Title: Comparison Between Oral Melatonin and Hydroxyzine in Pediatric Patients Undergoing Adenotonsillectomy
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Sarah Mohamed Aly Omar Mousa, Dr, Minia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 505/2022
Record Dates: First submitted 2022-12-19; First posted 2023-01-11 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Effect of Drug; Anxiety
Keywords: Melatonin; Hydroxyzine; Preoperative Anxiety; Pediatric; Adenotonsillectomy
MeSH Terms: conditions — Anxiety Disorders | interventions — Melatonin; Hydroxyzine

STUDY DESIGN:
Intervention Model Description: Three study groups
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Melatonin (Active Comparator): Preoperative oral melatonin 0.1mg/ kg in 10ml apple juice one hour before induction of anesthesia
  Interventions: Drug: Melatonin 3 MG
- Hydroxyzine (Active Comparator): Preoperative oral hydroxyzine 1mg/ kg in 10ml apple juice one hour before induction of anesthesia
  Interventions: Drug: Hydroxyzine Pill
- placebo (Placebo Comparator): 10ml apple juice one hour before induction of anesthesia
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Melatonin 3 MG — 0.1 mg/ kg melatonin in 10 ml apple juice 1 hour before induction of anesthesia
  Other Names: Melatonin
  Arms: Melatonin
Drug: Hydroxyzine Pill — 1 mg/ kg hydroxyzine in 10 ml apple juice 1 hour before induction of anesthesia
  Other Names: Atarax 10mg
  Arms: Hydroxyzine
Other: Placebo — 10 ml apple juice 1 hour before induction of anesthesia
  Arms: placebo

SUMMARY:
Comparison between the effect of oral Melatonin and Hydroxyzine for Preventing Preoperative Anxiety in pediatric Patients Undergoing Adenotonsillectomy

DETAILED DESCRIPTION:
The aim of the study is to compare the effectiveness of preoperative oral melatonin and hydroxyzine on preoperative anxiety in pediatric patients undergoing adenotonsillectomy.

The primary outcomes:

1. Ease of parenteral separation.
2. The compliance to anesthesia induction in pediatric patients.

The secondary outcomes:

1. Assessment of postoperative pain.
2. Time to first analgesic request.

ELIGIBILITY:
Inclusion Criteria:

1. ASA: class l
2. Sex: male and female
3. Age: from 3 to 10 years old
4. Children scheduled for adenotonsillectomy

Exclusion Criteria:

1. All children with a history of chronic illness, or developmental delay were excluded from the study
2. History of an autoimmune disease
3. Concurrent use of immunosuppressive treatment
4. Sleep disturbances, speech or communication problems
5. allergic to hydroxyzine, cetirizine, or other derivatives of piperazine, aminophylline, and ethylenediamine.
6. hydroxyzine is contraindicated in patients with acute porphyria

   -

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 78 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-01-30 (Estimated); Study Completion 2024-01-30 (Estimated)

PRIMARY OUTCOMES:
Ease of parenteral separation. | 20-30 minutes after administration
  Recorded as excellent, good, fair, or poor when the child is separated from the parent
The compliance to anesthesia induction in pediatric patients. | one hour after administration
  Assessed by a modified Yale preoperative anxiety scale, the range is from 5 to 22, the lower score is better

SECONDARY OUTCOMES:
Assessment of postoperative pain | immediately before and at induction procedure
  Face, Leg, Activity, Cry, and Consolability (FLACC) Scale from 0 to 10, the lower score is better
First analgesic request | Three hours postoperative
  Paracetamol

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Omar, Study Director — Minia University
Locations (1):
- Sarah Omar, Al Minyā, Egypt

IPD SHARING:
Plan to Share IPD: No
May share when the study is completed